CLINICAL TRIAL: NCT02016196
Title: Double Blind Randomized Study, Comparing Rifaximin vs Placebo for the Prevention of Encephalopathy in Patients Treated by TIPS
Brief Title: Rifaximin vs Placebo for the Prevention of Encephalopathy in Patients Treated by TIPS
Acronym: PRPET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/12/0551
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cirrhosis
Keywords: TIPS; portal pressure; rifaximin; overt hepatic encephalopathy; microbiota
MeSH Terms: conditions — Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rifaximin (Experimental): 6 rifaximin caps of 200 mg per day morning and night, during 15 days before TIPS, and after TIPS during 6 months.
  Interventions: Drug: Rifaximin
- placebo (Placebo Comparator): 6 caps placebo morning and night, 15 days before and 6 months after TIPS
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rifaximin — 6 rifaximin caps of 200 mg morning and night, 15 days before and 6 months after TIPS
  --------------------------------------------------------------------------------
  Other Names: NORMIX
  Arms: rifaximin
Drug: placebo — 6 placebo caps per day morning and night, during 15 days before TIPS and 6 months after TIPS
  Arms: placebo

SUMMARY:
TIPS has been used for 20 years, as a means of reducing portal pressure in patients with cirrhosis and portal hypertension related complications. TIPS proved more effective than alternative treatments in controlling or preventing variceal bleeding and refractory ascites. The main drawback of the TIPS procedure is progressive overt hepatic encephalopathy (OHE). Three risk factors for post-TIPS OHE have been identified: age over 65 years, history of previous episodes of OHE, and Child-Pugh score equal to or over 10. However, the incidence of post-TIPS OHE in patients fulfilling these criteria remains close to 35 %.

DETAILED DESCRIPTION:
TIPS has been used for 20 years, as a means of reducing portal pressure in patients with cirrhosis and portal hypertension related complications. TIPS proved more effective than alternative treatments in controlling or preventing variceal bleeding and refractory ascites. The main drawback of the TIPS procedure is progressive overt hepatic encephalopathy (OHE). Three risk factors for post-TIPS OHE have been identified: age over 65 years, history of previous episodes of OHE, and Child-Pugh score equal to or over 10. However, the incidence of post-TIPS OHE in patients fulfilling these criteria remains close to 35 %. Furthermore, the pathogenesis of HE in general but also in patients treated by TIPS is still not well understood. Therefore, there is a real challenge in discovering new molecular mechanisms involved in pathogenesis of OHE as well as new treatment to better prevent the risk of OHE in patients treated by TIPS. Observational and experimental studies suggest a microbiota's role in the mechanism of OHE and recently a non absorbable antibiotic has proven to reduce the risk of recurrence of OHE. However, the effect of this drug for the prevention of a first episode of OHE in patients treated by TIPS is not known. In addition, the mechanisms of the beneficial effect of rifaximin remain poorly understood.

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis with TIPS for ascit treatment or hydrothorax
* prevention digestive bleeding follow up portal hypertension -
* signed consent

Exclusion Criteria:

* hepatocellular carcinoma out of Milan criteria or palliative phase cancer
* Child Pugh score > 12
* TIPS indicated for other indication than bellow
* encephalopathy signs : asterixis or confusion
* Hypersensibility to rifaximin, or derivated of rifamycin
* Patients treated by same class antibacterial
* pregnant woman
* Patient with hepatic transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
First episode of overt encephalopathy in patients treated by TIPS | 6 months
  First episode of overt encephalopathy in patients treated by TIPS

SECONDARY OUTCOMES:
number of hospitalisation days | 6 months
  Number and days of hospitalisations for encephalopathy
Frequency of kidney insufficiency | 6 months
  number of digestive bleeding follow up to portal hypertension, number of ascit punctions, frequency kidney insufficiency and hepatocellular carcinoma
transplants, deaths | 6 months
  - number of transplants and deaths
intestinal microbiota | 6 months
  Composition of intestinal microbiota in 30 patients (only UHToulouse)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Bureau, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (13):
- France (13):
  - CHU Angers, Angers
  - Hôpital Jean Verdier, Bondy
  - CHU Bordeaux, Bordeaux
  - CHRU Lille, Lille
  - CHU Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU Beaujon Clichy, Paris
  - CHU Saint-Antoine, Paris
  - Pitié Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - UHToulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Bureau C, Thabut D, Jezequel C, Archambeaud I, D'Alteroche L, Dharancy S, Borentain P, Oberti F, Plessier A, De Ledinghen V, Ganne-Carrie N, Carbonell N, Rousseau V, Sommet A, Peron JM, Vinel JP. The Use of Rifaximin in the Prevention of Overt Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt : A Randomized Controlled Trial. Ann Intern Med. 2021 May;174(5):633-640. doi: 10.7326/M20-0202. Epub 2021 Feb 2. PMID 33524293